CLINICAL TRIAL: NCT05403398
Title: Change in Markers of Immune Function Associated With Bacillus Subtilis CU1 Intervention in Different Age Groups
Brief Title: BSCU1 and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lesaffre International (Industry)
Collaborators: NIZO Food Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL79890.000.21
Record Dates: First submitted 2022-05-20; First posted 2022-06-03 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2022-05

CONDITIONS: General Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BSCU1 (Experimental): B. subtilis CU1 at 2 billion CFUs daily for 4 weeks
  Interventions: Dietary Supplement: B. subtilis CU1

INTERVENTIONS:
Dietary Supplement: B. subtilis CU1 — 2 billion CFUs daily, for 4 weeks
  Other Names: B. subtilis CNCM I-2745

SUMMARY:
The current study aims to explore a range of possible pathways by which BSCU1 could beneficially modulate the immune system, in three target populations representing the general population.

DETAILED DESCRIPTION:
This exploratory study is designed as a single-arm study with repeated measures, involving three different populations, in which each subject serves as its own control. The duration of the intervention is 4 weeks, with biomarker assessments at baseline, after 2 weeks, and after 4 weeks intervention.

ELIGIBILITY:
Inclusion Criteria:

Adults

* 30 ≤ age ≤ 49 years
* BMI ≥ 18.5 and ≤ 25 kg/m2
* In good health as assessed during screening (by questionnaire), and the medical investigator's professional judgment
* Non-smoking

Elderly

* 65 ≤ age ≤ 79 years
* BMI ≥ 22.0 and ≤ 28.0 kg/m2
* Generally healthy as assessed during screening (by questionnaire), and the medical investigator's professional judgment
* Non-smoking

Children

* 3 ≤ age ≤ 6 years
* Healthy BMI, cut-off points will be used as indicated by JGZ
* Generally healthy as assessed during screening (by parental anamnesis), and the study physician's professional judgment

Exclusion Criteria:

Adults and elderly

* Chronic illness (e.g., diabetes mellitus, cardiac insufficiency, respiratory insufficiency, cancer, chronic kidney or liver disease),
* Acute infection in the past month
* Gastrointestinal disorders (e.g., inflammatory bowel disease),
* Acute gastroenteritis in the past 2 months
* Any vaccination in the past month or any scheduled vaccination during the study period
* Treatment with antibiotics within 2 months before the start of the study and during the study period
* Regular use of laxative agents
* Immunodeficiency disorder
* Use of anti-inflammatory or immunosuppressive drugs (e.g.cyclosporine, azathioprine, systemic corticosteroids, antibodies)
* Unexplained weight loss or weight gain of > 3 kg in the 3 months prior to pre-study screening
* Regular consumption of probiotics within 1 month before start of the study
* Evidence of current excessive alcohol consumption (>4 consumptions/day or >20 consumptions/week) or drug (ab)use
* Mental status that is incompatible with the proper conduct of the study

Children

* Acute respiratory or gastrointestinal infection in the past month
* Chronic illness (e.g. chronic infections, systemic or metabolic disease)
* Gastrointestinal disorders (e.g., inflammatory bowel disease),
* Acute gastroenteritis in the past 2 months
* Any vaccination in the past month or any scheduled vaccination during the study period
* Treatment with antibiotics within 2 months before the start of the study and during the study period
* Immunodeficiency disorder
* Use of anti-inflammatory or immunosuppressive drugs (e.g.cyclosporine, azathioprine, systemic corticosteroids, antibodies)
* Regular use of laxative agents
* Regular consumption of probiotics within 1 month before start of the study

Ages: 3 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Fecal sIgA | 4 weeks
  Change in fecal sIgA concentration

SECONDARY OUTCOMES:
Serum cytokine concentration | 4 weeks
  Change in serum cytokines concentration (e.g. MIP-1α, IL-6, Il-10, IFN-γ, TNF-α, IL-1β) in elderly using a commercial Multiplex Bead Immunoassay (Bio-Rad, Veenendaal, The Netherlands)
Ex-vivo cytokines concentration | 4 weeks
  Change in control and Lipopolysaccharide (LPS) stimulated cytokine (e.g. MIP-1α, IL-6, Il-10, IFN-γ, TNF-α, IL-1β) production in whole blood in adults and elderly using a commercial Multiplex Bead Immunoassay (Bio-Rad, Veenendaal, The Netherlands)
Ex-vivo phagocytosis | 4 weeks
  Ex-vivo phagocytic function of monocytes and granulocytes using the commercial pHrodo, BioParticles phagocytosis assay kit (Invitrogen, ThermoFisher) for flow cytometry
Fecal microbiota | 4 weeks
  Fecal microbiota composition using shotgun metagenomics sequencing
RNA sequencing | 4 weeks
  Gene expression in PBMC (RNA sequencing)
Immune cell phenotyping | 4 weeks
  Immune cell phenotyping will be performed by labelling of the cell with cell specific markers and measured by means of flow cytometry. Two panels of each 8-12 markers will be used for general cell phenotyping, including activation markers, and T cell specific phenotyping in PBMCs.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Jeanne, Study Director — Lesaffre Group
Locations (1):
- NIZO food research BV, Ede, ZB, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mourey F, Scholtens P, Jeanne JF, Rodriguez B, Decherf A, Machuron F, Kardinaal A, Scheithauer T, Porbahaie M, Narni-Mancinelli E, Crinier A. The probiotic strain Bacillus subtilis CU1 primes antimicrobial innate immune response and reduces low-grade inflammation: a clinical study. Benef Microbes. 2024 Aug 14;15(6):659-678. doi: 10.1163/18762891-bja00028. PMID 39151920